CLINICAL TRIAL: NCT06437613
Title: "Effects of Passive Static Stretching of 30 Seconds Versus 60 Seconds on the Hamstring Flexibility in Adults With Hamstring Tightness.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/9
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Hamstring Flexibility

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Week 1 Passive Hip Flexion Test Straight leg Raise Modified Knee Extension Test Passive Static Stretching 3-4 reps 3-5 second hold in each activity Week 2 Passive Hip Flexion Test Straight leg Raise Modified Knee Extension Test Passive Static Stretching 3-4 reps 3-5 second hold in each activity
  Week 3 Passive Hip Flexion Test Straight leg Raise Modified Knee Extension Test Passive Static Stretching 3-4 reps 3-5 second hold in each activity
  Week 4 Passive Hip Flexion Test Straight leg Raise Modified Knee Extension Test Passive Static Stretching 3-4 reps 3-5 second hold in each activity
  Interventions: Procedure: Passive Static Stretching exercises for 30 seconds
- Group 2 (Experimental): Week 1 Passive Hip Flexion Test Straight leg Raise Modified Knee Extension Test Passive Static Stretching 3-4 reps 3-5 second hold in each activity Week 2 Passive Hip Flexion Test Straight leg Raise Modified Knee Extension Test Passive Static Stretching 3-4 reps 3-5 second hold in each activity Week 3 Passive Hip Flexion Test Straight leg Raise Modified Knee Extension Test Passive Static Stretching 3-4 reps 3-5 second hold in each activity
  Week 4 Passive Hip Flexion Test Straight leg Raise Modified Knee Extension Test Passive Static Stretching 3-4 reps 3-5 second hold in each activity
  Interventions: Procedure: Passive Static Stretching exercises for 60 seconds

INTERVENTIONS:
Procedure: Passive Static Stretching exercises for 30 seconds — Intervention includes Following Tests
  1. Passive Hip Flexion Test(PHFT)
  2. Straight Leg Raises(SLR)
  3. Modified Knee Extension Test(MKET)
  Arms: Group 1
Procedure: Passive Static Stretching exercises for 60 seconds — Intervention includes Following Tests
  1. Passive Hip Flexion Test(PHFT)
  2. Straight Leg Raises(SLR)
  3. Modified Knee Extension Test(MKET)
  Arms: Group 2

SUMMARY:
This study is a randomised controlled trial and the purpose of this study is to determine the effects of Passive Static Stretching of 30 seconds versus 60 seconds on the Hamstring Flexibility in adults with Hamstring Tightness.

The study is conducted in Rehabilitation department of Fauji Foundation Hospital on the sample of 38 participants. Hamstring flexibility will be evaluated at the beginning by Active knee extension test.

The subjects will be randomized into two group by sealed envelope method. Baseline assessment would be done by using tools of SLR and modified knee extension test and then final assessment will be done after 4 weeks.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of passive static stretching on hamstring flexibility in adults with hamstring tightness" adults (age : 18-45 years ) by using

1. Goniometer
2. Straight leg raise (SLR)
3. Passive Hip Flexion Test(PHFT)
4. Active Knee Extension Test( AKET)
5. Modified Knee Extension Test(MKET) Data will be collected before and after the intervention protocol for each participant.

Data collection procedure:The subjects will be advised of the training session schedule following the baseline assessment. Pre and post intervention scores will be recorded.

ELIGIBILITY:
Inclusion criteria:

* Adults age ranging from 18-45 years
* Both males and females are included in the study
* Individuals with 90 degree hip flexion having a minimum reduction of 15 degrees in knee extension position.

Exclusion criteria :

* Old adults
* Individuals suffering from any acute or chronic co-morbidities of musculoskeletal, neurologic, cardiovascular or systemic origin
* Post-surgical cases
* Hamstring strain or any other dysfunction in past two years.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  Numeric Pain Rating Scale has a scale of 0-10 or 0-100 points and can be given verbally or in writing.
Range of motion | 4 weeks
  Goniometer will be used
Physical Function | 4 weeks
  Physical Function will be assessed using Oswestry disability Questionairre
Lumbar range of motion | 4 Weeks
  Using Inclinometer

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan